CLINICAL TRIAL: NCT00738075
Title: Online Automatic Recognition of Freezing of Gait Episodes
Brief Title: Automatic Recognition of Freezing of Gait Episodes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Nir Giladi MD, Tel Aviv Sourasky Medical Center
Other Study IDs: TASMC-08-NG-0283-CTIL
Record Dates: First submitted 2008-08-17; First posted 2008-08-20 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2008-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PD+FOG: Patients with Parkinson's disease prone to freezing
  Interventions: Device: Auditory cue

INTERVENTIONS:
Device: Auditory cue — When device recognizes automatically freezing episode it will generate auditory cue

SUMMARY:
The investigators hypothesize that mathematical algorithm can identify freezing episodes based on data obtained from accelerometer.

DETAILED DESCRIPTION:
The subjects will walk with an accelerometer. The acceleration traces will be online analyzed, and if freezing episode is recognized, an auditory cue will be heard.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinsons disease prone to freezing of gait

Exclusion Criteria:

* Patients who are not able to ambulate independently

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease prone to freezing of gait
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Meir Plotnik, PhD, Study Director — Tel-Aviv Sourasky Medical Center
Locations (1):
- Laboratory for Gait and Neurodynamics, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Moore ST, MacDougall HG, Ondo WG. Ambulatory monitoring of freezing of gait in Parkinson's disease. J Neurosci Methods. 2008 Jan 30;167(2):340-8. doi: 10.1016/j.jneumeth.2007.08.023. Epub 2007 Sep 2. PMID 17928063